CLINICAL TRIAL: NCT06851325
Title: Antiplatelets and Hemorrhagic MI
Brief Title: Antiplatelets and Intramyocardial Hemorrhage in STEMI: Incidence and Outcomes
Acronym: MIRON-PLATELET
Status: Completed | Type: Observational
Sponsor: Rohan Dharmakumar (Other)
Responsible Party: Sponsor-Investigator, Rohan Dharmakumar, Executive Director, Indiana University School of Medicine
Organization: Indiana University (Other)
Other Study IDs: 19978g
Record Dates: First submitted 2025-02-24; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: STEMI; Acute Myocardial Infarction
Keywords: Hemorrhagic Myocardial Infarction; Antiplatelets; MACE
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The MIRON-PLATELET study is a retrospective, observational multi-center analysis assessing the impact of different antiplatelet therapies on hemorrhagic myocardial infarction (HMI) incidence and outcomes in STEMI patients. Key endpoints include hemorrhagic transformation, MACE, bleeding complications, and 30-day mortality. Findings will offer insights into the safety and clinical implications of antiplatelet therapy in high-risk patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18-79 years at the time of STEMI diagnosis
2. Diagnosed with ST-segment elevation myocardial infarction (STEMI) based on standard clinical criteria
3. Received antiplatelet therapy as part of STEMI management
4. Underwent primary percutaneous coronary intervention (PCI)
5. Evidence of hemorrhagic MI confirmed by Cardiac Magnetic Resonance Imaging OR Post-PCI biomarker diagnostics
6. Availability of comprehensive medical records documenting STEMI presentation, treatment details, and clinical outcomes
7. Minimum of 30-day follow-up data, with extended follow-up available for up to 10 years

Exclusion Criteria:

1. Diagnosis of non-STEMI (NSTEMI), unstable angina, or other non-ischemic cardiomyopathies
2. History of prior hemorrhagic stroke or active intracranial bleeding before the index STEMI event
3. Known bleeding disorders (e.g., hemophilia, thrombocytopenia <50,000/µL)
4. Use of chronic antiplatelet therapy (aspirin, clopidogrel, ticagrelor, prasugrel) before STEMI diagnosis
5. Use of long-term anticoagulation therapy (warfarin, DOACs such as apixaban, rivaroxaban, dabigatran) before STEMI diagnosis
6. Incomplete or missing medical records preventing outcome assessment
7. History of malignancy with life expectancy <1 year at the time of STEMI diagnosis
8. Patients lost to follow-up before 30 days post-STEMI

Ages: 18 Years to 79 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients across multiple centers with available longitudinal follow-up data (up to 10 years), allowing for a comprehensive evaluation of clinical outcomes, mortality, major adverse cardiovascular events (MACE), and bleeding complications. Patients with a history of chronic antiplatelet or anticoagulation therapy before STEMI, known bleeding disorders, or incomplete medical records are excluded.
Sampling Method: Non-Probability Sample
Enrollment: 6180 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-02-11 (Actual)

PRIMARY OUTCOMES:
Incidence of Hemorrhagic Myocardial Infarction (HMI) in STEMI Patients Receiving Different Antiplatelet Therapies | 30 days post-STEMI diagnosis
  Risk ratio assessment of the occurrence of hemorrhagic transformation in STEMI patients treated with different antiplatelet regimens.

SECONDARY OUTCOMES:
Major Adverse Cardiovascular Events (MACE) | 10 years
  Composite of cardiovascular death, recurrent MI, stroke, and heart failure hospitalization.
Bleeding Complications | 10 years
  Incidence of major and minor bleeding events as per the BARC (Bleeding Academic Research Consortium) criteria.
All cause mortality | 10 years
  Evaluation of all-cause mortality at 30 days, 1 year, 5 years, and 10 years across different antiplatelet therapy groups.

CONTACTS AND LOCATIONS:
Overall Officials: Rohan Dharmakumar, PhD, Principal Investigator — Indiana University School of Medicine; Keyur P. Vora, MD FACC, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Krannert Cardiovascular Research Center, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vyas R, Changal KH, Bhuta S, Pasadyn V, Katterle K, Niedoba MJ, Vora K, Dharmakumar R, Gupta R. Impact of Intramyocardial Hemorrhage on Clinical Outcomes in ST-Elevation Myocardial Infarction: A Systematic Review and Meta-analysis. J Soc Cardiovasc Angiogr Interv. 2022 Aug 26;1(6):100444. doi: 10.1016/j.jscai.2022.100444. eCollection 2022 Nov-Dec. PMID 39132339
- [Background] Vora KP, Kumar A, Krishnam MS, Prato FS, Raman SV, Dharmakumar R. Microvascular Obstruction and Intramyocardial Hemorrhage in Reperfused Myocardial Infarctions: Pathophysiology and Clinical Insights From Imaging. JACC Cardiovasc Imaging. 2024 Jul;17(7):795-810. doi: 10.1016/j.jcmg.2024.02.003. Epub 2024 Apr 10. PMID 38613553